CLINICAL TRIAL: NCT02895334
Title: An Initial Evaluation of the MyHeartBaby Psychosocial Telemedicine Program
Brief Title: MyHeartBaby: An Initial Evaluation of the MyHeartBaby Psychosocial Telemedicine Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Pediatric Heart Network (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Brandon Aylward, Associate Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00082281
Record Dates: First submitted 2016-09-06; First posted 2016-09-09 (Estimated); Last update posted 2017-07-12 (Actual); Status verified 2017-07

CONDITIONS: Congenital Heart Disease
Keywords: CHD; Congenital Heart Disease
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- MyHeartBaby (Experimental): Caregivers will complete Telehealth Psychosocial Sessions and 4 follow up assessments.
  Interventions: Behavioral: MyHeartBaby Program
- Standard of Care (No Intervention): Caregivers will complete 4 follow up assessments.

INTERVENTIONS:
Behavioral: MyHeartBaby Program — Participating Caregivers will receive an electronic tablet loaded with a telemedicine intervention program (MyHeartBaby) to support caregivers remotely in the daily care and adjustment to having an infant with chronic medical needs with video-based telemedicine support services. There are a total of six sessions occurring at weeks 3, 6, 9, 12, and 15 of the study.
  Arms: MyHeartBaby

SUMMARY:
This study will conduct an initial clinical evaluation of this support program to examine its impact on reducing caregiver stress, increasing confidence in daily feeding, and improving weight-for-age growth percentiles in infants with Congenital Heart Disease (CHD).

DETAILED DESCRIPTION:
Caregivers of infants with CHD are at high-risk of anxiety and distress due to the complex daily caregiving demands. Previous research has demonstrated decreased parental stress and more optimal infant developmental outcomes with a psychosocial intervention delivered to caregivers of infants with CHD prior to hospital discharge as well as reduced healthcare use in caregivers who received medical video-consultations during the interstage surgical palliation period. This study will implement a telemedicine intervention program (MyHeartBaby) to support caregivers remotely in the daily care and adjustment to having an infant with chronic medical needs. The program is delivered via video chat over the Internet and caregivers will complete questionnaires about general family information, stress, and feeding their infant.

ELIGIBILITY:
Inclusion Criteria:

* Caregiver's infant is less than 45 days of age at time of study enrollment.
* Caregiver of infant with high-risk, shunt dependent physiology (one or two-ventricle circulation) having just received neonatal surgery for CHD.
* English is a primary language for caregiver of infant.

Exclusion Criteria:

* Caregiver's infant is greater than 45 days of age at time of study enrollment.
* Not a caregiver of infant with high-risk, shunt dependent physiology having just received neonatal surgery for CHD.
* English is not a primary language for caregiver of infant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2017-04-07 (Actual); Study Completion 2017-04-07 (Actual)

PRIMARY OUTCOMES:
Change in Levels Stress for Caregivers of 1-Ventricle Cardiac Defect Infants | Baseline, Week 18
  Stress levels will be measured by the Pediatric Inventory for Parents (PIP) which is a 42-item measure that assesses disease-related parenting stress and asks caregivers to indicate the frequency at which disease-related parenting stressor occurs, and the difficulty-level of each stressor.
Change in Levels Stress for Caregivers of 2-Ventricle Cardiac Defect Infants | Baseline, Week 18
  Stress levels will be measured by the Pediatric Inventory for Parents (PIP) which is a 42-item measure that assesses disease-related parenting stress and asks caregivers to indicate the frequency at which disease-related parenting stressor occurs, and the difficulty-level of each stressor.

SECONDARY OUTCOMES:
Change in Levels of Caregiver Confidence in Feeding Management for 1-Ventricle Cardiac Defect Infants | Baseline, Week 18
  The confidences in feeding questionnaire has been developed for purposes of this study and has a list of 20 questions that ask caregivers about daily feeding practices, stress associated with feeding, and ability to soothe infant.
Change in Levels of Caregiver Confidence in Feeding Management for 2-Ventricle Cardiac Defect Infants | Baseline, Week 18
  The confidences in feeding questionnaire has been developed for purposes of this study and has a list of 20 questions that ask caregivers about daily feeding practices, stress associated with feeding, and ability to soothe infant.
Change in Infant Weight for 1-Ventricle Cardiac Defect Infants | Baseline, Week 18
  Clinical assessments of weight-for-age percentiles for purposes of study outcomes will be obtained during regularly scheduled clinic visits.
Change in Infant Weight for 2-Ventricle Cardiac Defect Infants | Baseline, Week 18
  Clinical assessments of weight-for-age percentiles for purposes of study outcomes will be obtained during regularly scheduled clinic visits.
Number of Unplanned Hospital Admissions | Week 18
  Caregivers will report infant hospital admissions during the study duration.

CONTACTS AND LOCATIONS:
Overall Officials: Brandon Aylward, Principal Investigator — Emory University
Locations (1):
- Children's Healthcare of Atlanta, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No